CLINICAL TRIAL: NCT06260241
Title: Gain in Stretched Penile Length After Phalloplasty With & Without Penile Traction in Children.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shaikh Zayed Hospital, Lahore (Other)
Responsible Party: Principal Investigator, ADEEL AHMED, POST GRADUATE RESIDENT, Shaikh Zayed Hospital, Lahore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: ShaikhZayedH
Record Dates: First submitted 2023-12-11; First posted 2024-02-15 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Concealed Penis

STUDY DESIGN:
Intervention Model Description: Randomized Control Trial
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- With Traction Dressing (Other): Traction dressing will be applied to patients after phalloplasty for 24 hours.
  Interventions: Procedure: Traction Dressing
- Without Traction Dressing (Other): No traction dressing will be applied to patients after phalloplasty for 24 hours.
  Interventions: Other: Without Traction Dressing

INTERVENTIONS:
Procedure: Traction Dressing — Traction dressing will be applied to one group for 24 hours and simple dressing to the other group.
  Arms: With Traction Dressing
Other: Without Traction Dressing — Without Traction Dressing
  Arms: Without Traction Dressing

SUMMARY:
The goal of this Randomized Controlled Trial is to assess the gain in stretched penile length after phalloplasty with & without penile traction in children of age group 4 to 13 years presenting in hospital with the complaint of concealed penis.

The main question[s] it aims to answer is:

• Gain in stretched penile length after phalloplasty with and without penile traction in children.

DETAILED DESCRIPTION:
Concealed penis is a rare clinical entity that affects young males. It leads to various concerns about cosmesis even though it does not necessarily affect functional aspects such as micturition and intercourse. However, data suggests that up to 4% of individuals may be affected by a concealed penis and this can lead to great distress to the patient especially as the child ages. There are different methods of phalloplasty that are performed, however none have explored the possible benefit of traction to the penis after phalloplasty to increase stretched penile length. We conducted a pilot study where we found a modest increase in stretched penile length following traction with phalloplasty and believe that addition of this step will help individuals with a concealed penis following phalloplasty gain a modest increase in length. The hypothesis of this study is that there will be a significant mean gain in stretched penile length with traction for 24 hours following phalloplasty for concealed penis. The research conducted will be a Randomized Control Trial with two groups where one group receives traction while one group does not.

The net gain in stretched penile length, stretched penile length pre-operatively and 2 weeks post-operatively will be analyzed using the independent study T-test with a P-value of 0.05 or less as significant between the two groups. The difference between the baseline SPL and post-operative SPL for each group will be assessed using the paired student t-test with a p-value less than 0.05 as significant. Sample Size for our study will be 70 patients (35 in each group).

Phalloplasty is a well-known procedure in children presenting with concealed penis as ordinary circumcision may lead to phimosis and adhesions formation between glans and skin in concealed penis. This procedure is not associated with any untoward results (except Suture Cut-through the glans skin which can be easily repaired) as only traction will be applied & SPL will be measured immediately per-op & two weeks post operatively.

Since there is currently no local study assessing the increase in stretched penile length following phalloplasty with traction, we have done a pilot study (Annexure B) whose results were satisfactory with penile traction as compared to without penile traction therefore, we anticipate a notable augmentation in stretched penile length both prior to and post the procedure in each patient. This observation implies that employing 24-hour penile traction may be a recommended course of action, potentially opening the door for more comprehensive investigations to furnish additional evidence regarding the procedure's advantages. It is important to acknowledge that this study will face limitations due to the restricted sample size, primarily attributable to the rare nature of the condition. Given the limited existing literature on the subject, the substantial prevalence of the condition, and the absence of a consensus regarding the optimal approach for concealed penis, this study could contribute to the existing body of knowledge by examining the efficacy of combining penile traction with phalloplasty.

ELIGIBILITY:
Inclusion Criteria:

* Infants and children aged 4 years to 13 years of age.
* Presenting with concealed penis for circumcision.

Exclusion Criteria:

* Congenital Buried Penis
* Webbed penis
* Structural abnormalities of the penis such as hypospadias, Epispadias etc.
* Existing co-morbid syndromes or conditions
* Unfit for general anesthesia
* Known bleeding diathesis
* Incomplete foreskin
* Any previous penile surgery

Ages: 4 Years to 13 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — Male
Enrollment: 70 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
The gain in stretched penile length (SPL) | up to 2 Years
  To measure the gain in stretched penile length (SPL) following phalloplasty with and without penile traction applied for 24 hours for patients undergoing surgery for concealed penis at two weeks post-operatively.

CONTACTS AND LOCATIONS:
Overall Officials: MUHAMMAD ALI SHEIKH, MBBS FCPS, Study Chair — SHEIKH ZAYED HOSPITAL
Locations (1):
- Sheikh Zayed Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Brisson P, Patel H, Chan M, Feins N. Penoplasty for buried penis in children: report of 50 cases. J Pediatr Surg. 2001 Mar;36(3):421-5. doi: 10.1053/jpsu.2001.21605. PMID 11226987
- [Result] Hadidi AT. Buried penis: classification surgical approach. J Pediatr Surg. 2014 Feb;49(2):374-9. doi: 10.1016/j.jpedsurg.2013.09.066. Epub 2013 Nov 7. PMID 24528990
- [Result] Hampson LA, Muncey W, Chung PH, Ma CC, Friedrich J, Wessells H, Voelzke BB. Surgical and Functional Outcomes Following Buried Penis Repair With Limited Panniculectomy and Split-thickness Skin Graft. Urology. 2017 Dec;110:234-238. doi: 10.1016/j.urology.2017.07.021. Epub 2017 Aug 7. PMID 28797684
- [Result] Heston AL, Esmonde NO, Dugi DD 3rd, Berli JU. Phalloplasty: techniques and outcomes. Transl Androl Urol. 2019 Jun;8(3):254-265. doi: 10.21037/tau.2019.05.05. PMID 31380232
- [Result] Ho TS, Gelman J. Evaluation and management of adult acquired buried penis. Transl Androl Urol. 2018 Aug;7(4):618-627. doi: 10.21037/tau.2018.05.06. PMID 30211051